CLINICAL TRIAL: NCT01752413
Title: Iron Depletion and Replacement in Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Blood Centers, Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IDAR-PN
Record Dates: First submitted 2012-12-10; First posted 2012-12-19 (Estimated); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Anemia
Keywords: Iron depletion; blood donors; iron replacement
MeSH Terms: conditions — Anemia | interventions — ferrous gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferrous gluconate 325mg (Experimental): Those found iron depleted by ferritin measure will receive 325 mg Ferrous gluconate twice a day for 100 days. They will be deferred as a whole blood donor for 120 days until completion of iron therapy. They will receive standard dietary counseling.
  Interventions: Dietary Supplement: Ferrous gluconate 325mg; Behavioral: Nutrition counseling
- Nutrition counseling (Active Comparator): For those consenting to this study but who demonstrate adequate ferritin levels (>20 micrograms/L female, >30 micrograms/L males), they will not receive oral iron or additional deferral period but will be allowed to donate after the standard 56 days. They will receive standard counseling about iron rich foods. Rate and frequency of subsequent donations will be tracked and compared to those receiving iron supplementation.
  Interventions: Behavioral: Nutrition counseling

INTERVENTIONS:
Dietary Supplement: Ferrous gluconate 325mg — Participants with low ferritin (<30 micrograms/L (males) or <20 micrograms/L (females)) will be asked to take two tablets of Ferrous Gluconate 325 mg (36 mg elemental iron) per day.
  Arms: Ferrous gluconate 325mg
Behavioral: Nutrition counseling — All blood donors receive current dietary counseling recommending iron rich foods

SUMMARY:
The purpose of this study is to determine (1) the role of ferritin testing to screen for iron depletion in donors at risk of low iron levels (2) the effectiveness of oral iron replacement therapy on the repletion of iron stores in donors, and (3) the feasibility of blood centers to routinely distribute oral iron replacement therapy to donors.

DETAILED DESCRIPTION:
This prospective study will be conducted under IRB approval at Memorial Blood Centers. Approximately 1000 donors will be enrolled over a two-year period.

Participant Recruitment Donors presenting to donate whole blood at MBC who have a Hb value between 12.5-13.5 (males) or 12.0-13.0 (females) will be asked to participate. Written informed consent will be obtained from each participant.

STUDY PROCEDURES MBC will be responsible for donor consenting, specimen collection and testing, donor deferral, donor-follow-up, and record keeping. Before any study participation, donors who meet the inclusion criteria will be required to sign and date an informed consent. All participants will receive a study information sheet and be asked screening questions and donor information.

An EDTA and red top tube will be taken from the diversion pouch of each participant during their donation, or obtained from samples already drawn for donor screening. The EDTA sample and red top tube will be used to determine baseline CBC and ferritin levels, respectively.

Female participants who have a Hb of 12.0-12.4 will not be allowed to donate per FDA regulations, but will be asked to have an EDTA and red top tube drawn to determine baseline CBC and ferritin levels, respectively.

Participants whose ferritin levels are <30 (males) or <20 (females) will be eligible for enrollment into the low ferritin group. Those with ferritin levels >30 (males) or >20 (females) will be enrolled into the low Hb only group. Females whose Hb was in the range of 12.0-12.4 and with ferritin levels >20 will not be followed.

Once ferritin levels are determined, participants in both groups will be contacted by a study nurse. Those in the low Hb only group will be notified of their results and allowed to return after a standard 56 day deferral. Those in the low ferritin group will be offered iron replacement therapy and deferred from blood donation for 112 days.

Oral Iron Replacement Therapy Participants in the low ferritin group will be offered 200 tablets of Ferrous gluconate 325 mg (36 mg elemental iron) sent by mail. Tablets will be in child proof containers. This amount and form of iron were chosen because of its ready accessibility over the counter in packs of 100 at low cost to donor/donor center. Also, the following anemia website suggests 60mg elemental iron daily, i.e. 2-3 iron tablets in divided doses daily.Participants will be instructed to take one at lunch and one at bedtime. Participants will be instructed to contact the study physician or study nurse immediately if any adverse events occur.

Between 25 and 35 days, the study physician or nurse will contact all participants in the low ferritin group to assess their compliance and tolerance with the iron replacement therapy using a standard instrument. Those with unacceptable intolerance to the ferrous gluconate may be offered carbonyl iron at this time, and re-interviewed between days 60 and 70 using the same instrument.

Participant Follow-Up Participants in both groups will be asked to return to donate after their deferral period. During their follow-up donation, participants will be asked to complete a follow-up questionnaire, and samples will again be taken to determine CBC and ferritin levels. Participants will be notified of their results. Statistical analysis will be performed to determine outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Fingerstick Hb value of 12.5-13.5 (males) or 12.0-13.0 (females)
* Meets all other blood donor inclusion criteria
* =>18 years of age

Exclusion Criteria:

* History or family history of hemochromatosis, colon cancer, intestinal polyps, or chronic gastrointestinal disease
* Currently taking iron in a form other than a multivitamin
* Currently on a chronic therapeutic use of NSAIDS or anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed B. Gorlin, MD, MBA, Principal Investigator — Memorial Blood Centers
Locations (1):
- Memorial Blood Centers, Saint Paul, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferrous Gluconate 325mg | Nutrition Counseling
Started | 170 | 27
Completed | 58 | 6
Not Completed | 112 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferrous Gluconate 325mg | Nutrition Counseling | Total
Number analyzed (Participants) | 170 | 27 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 128 | 23 | 151
  >=65 years | 41 | 4 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 17 | 147
  Male | 40 | 10 | 50
Region of Enrollment [Number; unit: participants]
  United States | 170 | 27 | 197

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adherence to Iron Replacement Therapy at Subsequent Donation
Description: Subject self reported habits for taking iron supplement or iron rich diet and severity of gastrointestinal complaints (minimal-1 to severe-5). GI complaints were not separated by type for analysis.
Time Frame: Two years
Population: Repeat Blood Donors
Measure: Count of Participants; unit: Participants
Arm/Group | Ferrous Gluconate 325mg | Nutrition Counseling
Number analyzed (Participants) | 170 | 27
Participants | 116 | 17

2. Secondary Outcome: Number of Participants With Improved Ferritin Levels on Subsequent Visit
Description: Compared ferritin levels at baseline and after iron replacement therapy among blood donors, adjusting for time between visits, participant adherence levels, and whether a unit was donated at second visit.
Time Frame: Two years
Measure: Count of Participants; unit: Participants
Arm/Group | Ferrous Gluconate 325mg | Nutrition Counseling
Number analyzed (Participants) | 116 | 17
Participants | 73 | 6

ADVERSE EVENTS:
Time Frame: Two Years post initial donation
Description: Gastrointestinal complaints self reported by subject on a scale of 1 for Minimal to 5 for Severe. Complaints grouped for analysis.
Arm/Group | Ferrous Gluconate 325mg | Nutrition Counseling
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/27
Other Adverse Events (participants affected / at risk) | 35/170 | 6/27
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferrous Gluconate 325mg (N=170) | Nutrition Counseling (N=27)
GI complaints (Gastrointestinal disorders) | 35 (35) | 6 (6) — diarrhea/constipation/dark stools

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes